CLINICAL TRIAL: NCT03189082
Title: "Microbotox" Versus Intramuscular Botulinum Toxin in Lower Face Rejuvenation: A Crossover Clinical Trial
Brief Title: Microbotox for Lower Face Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, samer jabbour, M.D., St Joseph University, Beirut, Lebanon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USJ-04
Record Dates: First submitted 2017-06-09; First posted 2017-06-16 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Botulinum Toxin; Rejuvenation; Therapy; Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Procedure: Microbotox

INTERVENTIONS:
Procedure: Microbotox — Microbotox is the injection of multiple microdroplets of diluted botulinum toxin into the dermis of the lower face

SUMMARY:
The purpose of this study is to evaluate the efficiency of the intradermal injection of botulinum toxin in lower face rejuvenation. The study will also compare this intervention with the "Nefertiti Lift" intramuscular injection technique.

DETAILED DESCRIPTION:
The abobotulinumtoxinA will be used for the intervention. The abobotulinumtoxinA will be prepared by adding 2.5 cc of normal saline to a 500-unit Dysport© (Ipsen Ltd, Berks, UK) vial. Further dilution to the appropriate Microbotox concentration will be done in the syringe itself. Each 1mL syringe of Microbotox solution will contain 20-28 units of onabotulinumtoxinA per mL of solution.

Preinjection frontal, oblique and lateral patient pictures will be taken (at rest and with contraction)

Injection points:

A series of 100-150 intradermal microdroplets injection points 1 cm apart will be delivered in the lower face. The area to be injected is bounded by a line 3 fingerbreadths above and parallel to the lower border of the mandible, 1 fingerbreadth posterior to the depressor anguli oris, and all the way down over the cervicomental angle and anterior neck to the upper border of the clavicle, and posteriorly to the anterior border of the sternocleidomastoid.

In the average patient, 2 syringes of 28 units per mL of microbotox will be used to cover the entire area.

In heavier necks, 3 syringes of 28 units per mL will be used. In thinner necks, 2 syringes of 20 units per mL will be used.

Follow up will be done at 15 days for post injection pictures. A total of 15 patients will be recruited

ELIGIBILITY:
Inclusion Criteria:

Female patients presenting to our clinic for neck rejuvenation who:

* Were deemed nonsurgical candidates for neck rejuvenation
* Were not willing to undergo invasive surgical procedures
* Had a medical contraindication to surgery

Exclusion Criteria:

* Patients with lower face botulinum toxin injection in the past 12 months
* Patients with resorbable lower face fillers injection in the past 12 months
* Patients with previous permanent lower face fillers injection
* Pregnant patients
* Lactating patients
* Patients with preexisting neuromuscular conditions (myasthenia gravis, Eaton Lambert syndrome)
* Patients using medication that could potentiate the effect of botulinum (ex: aminoglycoside antibiotics)
* Patients with sensitivity to botulinum toxin or human albumin

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Neck volume using a validated scale from the Summit Scale II | 15-25 days post treatment
  The assessment will be done by 3 plastic surgeons. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale. The 3 evaluators will be blinded to the pre or post injection status of the photos.
  1. No Sagging
  2. Mild Sagging
  3. Moderate Sagging
  4. Severe Sagging
  5. Very Severe Sagging
Jowls at rest using a validated scale from the Summit Scale II | 15-25 days post treatment
  The assessment will be done by 3 plastic surgeons. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale. The 3 evaluators will be blinded to the pre or post injection status of the photos
  1. No Sagging
  2. Mild Sagging
  3. Moderate Sagging
  4. Severe Sagging
  5. Very Severe Sagging
Marionette lines at rest using a validated scale from the Summit Scale II | 15-25 days post treatment
  The assessment will be done by 3 plastic surgeons. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale. The 3 evaluators will be blinded to the pre or post injection status of the photos
  1. No visible folds: continuous skin lines
  2. Shallow but visible folds with slight indentation
  3. Moderately deep folds, clear feature at normal appearance, but not when stretched
  4. Very long and deep folds, prominent facial feature
  5. Extremely long and deep folds; detrimental facial appearance
Oral commissures at rest using a validated scale from the Summit Scale II | 15-25 days post treatment
  The assessment will be done by 3 plastic surgeons. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale. The 3 evaluators will be blinded to the pre or post injection status of the photos
  1. No Downturn
  2. Mild Downturn
  3. Moderate Downturn
  4. Severe Downturn
  5. Very Severe Downturn
Platysmal bands at maximal contraction using a validated scale | 15-25 days post treatment
  The assessment will be done by 3 plastic surgeons. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale. The 3 evaluators will be blinded to the pre or post injection status of the photos
  1. No relevant prominence of platysmal bands
  2. Mild prominence of platysmal bands
  3. Moderate prominence of platysmal bands
  4. Severe prominence of platysmal bands
  5. Very severe prominence of platysmal bands
Platysmal bands at rest using a validated scale | 15-25 days post treatment
  The assessment will be done by 3 plastic surgeons. Pre and post injection scores will be calculated by the independent evaluators based on the photographic scale.
  1. No platsymal bands visible at rest
  2. Mild platysmal bands evident at rest. Bands do not appear along the full length of the neck.
  3. Mild platysmal bands evident along the full length of the neck at rest, less than 5 mm of elevation from the surrounding tissue.
  4. Moderate platsymal bandsvisible at rest along the full length of the neck, elevation at least 5 mm from the surrounding tissue.
  5. Severe platsymal bands along the full length of the neck at rest, elevation at least 5 mm from the surrounding tissue, with additional soft tissue ptotic banding present laterally
Mandibular definition change with maximal contraction will be assessed by a 2-point scale | 15-25 days post treatment
  The assessment of the pre-injection photos will be done by 3 plastic surgeons.
  1. Mandibular contour does not worsen with platysmal contraction
  2. Mandibular contour worsen with platysmal contraction

SECONDARY OUTCOMES:
Investigators Global Aesthetic Improvement Scale | 15-25 days post treatment
  Improvement in Overall appearance (global neck, jowls, skin laxity, platysmal bands, mandibular contour), as assessed by the investigators using the Global Aesthetic Improvement Scale (GAIS). GAIS will be completed based on photographic assessment comparing post-treatment photos taken at day 15-25 post intervention to baseline photos, to assess overall aesthetic improvement. The GAIS is a 5-point scale (1-5) as follows:
  1. Very Much Improved: optimal cosmetic results
  2. Much Improved: marked improvement in appearance from initial condition but not completely optimal
  3. Improved: obvious improvement in appearance from initial condition but additional treatments are advised
  4. No Change: the appearance is the same as the original condition
  5. Worse: the appearance is worse from the original condition
Subject Global Aesthetic Improvement Scale | 15-25 days post treatment
  Improvement in Overall appearance (global neck, jowls, skin laxity, platysmal bands, mandibular contour), as assessed by the subject using the Global Aesthetic Improvement Scale (GAIS). GAIS will be completed based on a live assessment of the subject with a mirror in hand for real time assessment and and a photographic assessment comparing post-treatment photos taken at day 15-25 post intervention to baseline photos, to assess overall aesthetic improvement. The GAIS is a 5-point scale (1-5) as follows:
  1. Very Much Improved: optimal cosmetic results
  2. Much Improved: marked improvement in appearance from initial condition but not completely optimal
  3. Improved: obvious improvement in appearance from initial condition but additional treatments are advised
  4. No Change: the appearance is the same as the original condition
  5. Worse: the appearance is worse from the original condition
Patient satisfaction | 15-25 days post treatment
  Patient satisfaction will be determined by a questionnaire completed at 15-25 days post-treatment. Subjects will indicate how satisfied they are on a 4-point scale (1-4) as follow:
  1. Very Satisfied
  2. Satisfied
  3. Dissatisfied
  4. Very Dissatisfied.
Patient willingness to repeat the procedure | 15-25 days post treatment
  Patient willingness to repeat the procedure will be assessed by a simple question with a Yes or No response
Patient willingness to recommend the procedure | 15-25 days post treatment
  Patient willingness to recommend the procedure to a friend will be assessed by a simple question with a Yes or No response
Assessment of Pain during treatment | Immediately after the treatment
  Subjects' pain during the treatment will be recorded using a validated Numeric Rating Scale (0-10), with 0 representing no pain and 10 representing the worst pain possible

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Dieu De France, Beirut, Aschrafieh, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Awaida CJ, Jabbour SF, Rayess YA, El Khoury JS, Kechichian EG, Nasr MW. Evaluation of the Microbotox Technique: An Algorithmic Approach for Lower Face and Neck Rejuvenation and a Crossover Clinical Trial. Plast Reconstr Surg. 2018 Sep;142(3):640-649. doi: 10.1097/PRS.0000000000004695. PMID 29879010